CLINICAL TRIAL: NCT01430429
Title: An Open Label Single Arm Study to Investigate the Safety and Efficacy of Multiple Administrations of NI-0801, a Fully Human Anti-CXCL10 Monoclonal Antibody in PBC Patients With an Incomplete Response to Ursodeoxycholic Acid
Brief Title: Primary Biliary Cirrhosis: Investigating A New Treatment Option Using NI-0801, an Anti-CXCL10 Monoclonal Antibody
Acronym: PIANO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Light Chain Bioscience - Novimmune SA (Industry)
Responsible Party: Sponsor
Other Study IDs: NI-0801-03
Record Dates: First submitted 2011-09-05; First posted 2011-09-08 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2012-06

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NI-0801 (Experimental)
  Interventions: Drug: NI-0801

INTERVENTIONS:
Drug: NI-0801

SUMMARY:
The purpose of the study is to assess safety and efficacy of multiple doses of NI-0801 in primary biliary cirrhosis patients with an inadequate response to ursodeoxycholic acid.

ELIGIBILITY:
Inclusion Criteria:

* Proven primary biliary cirrhosis (PBC), as demonstrated by the presence of at least 2 of the following 3 diagnostic factor (History of increased alkaline phosphatase levels for at least 6 months; positive serum AMA titer; Liver biopsy consistent with PBC)
* Elevated liver enzyme levels at screening
* Have given written informed consent

Exclusion Criteria:

* Screening bilirubin > 2.9 mg/dL (50 μmol/L)
* Screening creatinine clearance < 80 ml/min
* History or presence of hepatic decompensation (e.g., esophageal variceal bleeding, hepatic encephalopathy, or ascites)
* Positive serology result for Human Immunodeficiency Virus (HIV), Hepatitis B or C
* Known or previous diagnosis of malignancy
* Presence of any active infection
* Previous history of active TB within 12 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- IRCCS Istituto Clinico Humanitas, Rozzano, Italy
- NIHR Liver Biomedical Research Unit, Queen Elizabeth Hospital, Birmingham, United Kingdom

REFERENCES:
- [Derived] Mousa HS, Lleo A, Invernizzi P, Bowlus CL, Gershwin ME. Advances in pharmacotherapy for primary biliary cirrhosis. Expert Opin Pharmacother. 2015 Apr;16(5):633-43. doi: 10.1517/14656566.2015.998650. Epub 2014 Dec 29. PMID 25543678